CLINICAL TRIAL: NCT01745471
Title: Adipose Tissue Angiogenesis in Polycystic Ovary Syndrome (PCOS)
Brief Title: Adipose Tissue and Polycystic Ovary Syndrome (PCOS)(EIFFEL)
Acronym: EIFFEL
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Sanford-Burnham Medical Research Institute (Other); Pennington Biomedical Research Center (Other); Boston University (Other); Tufts University (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMDFH 348525; 348525 (Other: AdventHealth)
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome; Metabolic Diseases; Overweight
Keywords: Abdominal Adipose; Gluteal Adipose; Polycystic Ovary Syndrome; Obesity; Women
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Diseases; Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine Adipose tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PCOS group: 12 women with Polycystic Ovary Syndrome (PCOS) as defined by NIH criteria
- Pear shapes: 12 with an android pattern as defined by a waist-to-hip greater than 0.85
- Apple shapes: 12 will have a gynoid pattern as defined by a waist-to-hip ratio less than 0.78

SUMMARY:
The purpose of this study is to collect data to help understand why some women develop Polycystic Ovary Syndrome (PCOS) associated with decreased lower-body fat.

DETAILED DESCRIPTION:
Epigenetics may represent a new regulator mechanism explaining gluteal vs. abdominal fat differences.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 20 and < 40
* Weight stable (change of less than 3 kg in the last 8 weeks)
* BMI < 40 kg/m2 or > 27 kg/m2

Supplemental inclusion criteria for PCOS women:

* NIH criteria - confirmed by subjects' medical records.

Exclusion Criteria:

* Male
* Women who are pregnant or lactating (breast feeding)
* Post-menopausal women
* Women with hysterectomy
* Diagnosed with diabetes, or have a fasting blood sugar > 126 mg/dL.
* Untreated or symptomatic thyroid disease.
* Impaired kidney or liver function, as evidenced by your blood work
* Hypertension/ high blood pressure or are taking blood pressure medications
* Use of oral contraceptives or hormone replacement therapy.
* History of drug or alcohol abuse (> 3 drinks per day) in the last 5 years, or psychiatric disease prohibiting adherence to study protocol.
* History of cancer within the last 5 years.
* History of organ transplant.
* History of HIV, active Hepatitis B or C, or Tuberculosis.
* History of heart attack/ myocardial infarction.
* Presence of clinically significant abnormalities on EKG.
* Current smokers (smoking within the past 3 months)
* Use of any medications known to influence glucose, fat and/or energy metabolism within the last 3 months (e.g., growth hormone therapy, glucocorticoids [steroids], etc.). Metformin for women with PCOS is allowed.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population and screening: Healthy young women with a BMI > 30 will be recruited; 12 will have a gynoid pattern as defined by a waist-to-hip ratio less than 0.78 and 12 with an android pattern as defined by a waist-to-hip greater than 0.85. A third group will include 12 women with PCOS as defined by the NIH criteria. Subjects will be recruited via a dedicated website, physician referrals, direct mail outs, newspaper advertisements, and brochures. Only subjects that will sign informed consent and meet eligibility criteria will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2012-12-06 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference of angiogenesis capacity in abdominal and gluteal adipose tissue | Day 7
  The angiogenesis capacity of each adipose tissue depot will be determine by an in vitro angiogenesis test.

SECONDARY OUTCOMES:
Presence of biomarkers in abdominal and gluteal adipose tissue in obese and PCOS women | Day 7
  Measurement will be obtained with Fluorescence-activated cell sorting (FACS).
  Identify different and similar biomarkers in obese and PCOS women, from abdominal and gluteal adipose tissue samples. Total RNA, micro RNA and DNA will be extracted from each type of cells using FACS-cell sorting analysis.
Difference in oxygen content of abdominal and gluteal adipose tissue | Day 6
  Adipose tissue oxygen content will be measured using the Licox CMP microprocessor.

OTHER OUTCOMES:
The rates of carbohydrate oxidation | Day -7
  Resting Metabolic Rate (RMR) will measure the resting metabolic rate/respiratory quotient (RMR/RQ) and substrate utilization.
  Energy expenditure and respiratory quotient standardized for temperature, pressure, and moisture will be calculated at one-minute intervals, over 30 minutes.
The rates of lipid oxidation | Day -7
  Resting Metabolic Rate (RMR) will measure the resting metabolic rate/respiratory quotient (RMR/RQ) and substrate utilization.
  Energy expenditure and respiratory quotient standardized for temperature, pressure, and moisture will be calculated at one-minute intervals, over 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Divoux, PhD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes; Steven R Smith, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499
- [Background] Weber RV, Buckley MC, Fried SK, Kral JG. Subcutaneous lipectomy causes a metabolic syndrome in hamsters. Am J Physiol Regul Integr Comp Physiol. 2000 Sep;279(3):R936-43. doi: 10.1152/ajpregu.2000.279.3.R936. PMID 10956251
- [Background] Tran TT, Yamamoto Y, Gesta S, Kahn CR. Beneficial effects of subcutaneous fat transplantation on metabolism. Cell Metab. 2008 May;7(5):410-20. doi: 10.1016/j.cmet.2008.04.004. PMID 18460332
- [Background] Elbers JM, Asscheman H, Seidell JC, Megens JA, Gooren LJ. Long-term testosterone administration increases visceral fat in female to male transsexuals. J Clin Endocrinol Metab. 1997 Jul;82(7):2044-7. doi: 10.1210/jcem.82.7.4078. PMID 9215270
- [Background] Elbers JM, Asscheman H, Seidell JC, Gooren LJ. Effects of sex steroid hormones on regional fat depots as assessed by magnetic resonance imaging in transsexuals. Am J Physiol. 1999 Feb;276(2):E317-25. doi: 10.1152/ajpendo.1999.276.2.E317. PMID 9950792
- [Background] Shi H, Seeley RJ, Clegg DJ. Sexual differences in the control of energy homeostasis. Front Neuroendocrinol. 2009 Aug;30(3):396-404. doi: 10.1016/j.yfrne.2009.03.004. Epub 2009 Mar 31. PMID 19341761
- [Background] Perrot-Sinal TS. Do these genes make me look fat? Endocrinology. 2009 Mar;150(3):1075-7. doi: 10.1210/en.2008-1586. No abstract available. PMID 19240263
- [Background] Lavebratt C, Almgren M, Ekstrom TJ. Epigenetic regulation in obesity. Int J Obes (Lond). 2012 Jun;36(6):757-65. doi: 10.1038/ijo.2011.178. Epub 2011 Sep 13. PMID 21912396
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Cinti S, Mitchell G, Barbatelli G, Murano I, Ceresi E, Faloia E, Wang S, Fortier M, Greenberg AS, Obin MS. Adipocyte death defines macrophage localization and function in adipose tissue of obese mice and humans. J Lipid Res. 2005 Nov;46(11):2347-55. doi: 10.1194/jlr.M500294-JLR200. Epub 2005 Sep 8. PMID 16150820
- [Background] Strissel KJ, Stancheva Z, Miyoshi H, Perfield JW 2nd, DeFuria J, Jick Z, Greenberg AS, Obin MS. Adipocyte death, adipose tissue remodeling, and obesity complications. Diabetes. 2007 Dec;56(12):2910-8. doi: 10.2337/db07-0767. Epub 2007 Sep 11. PMID 17848624
- [Background] Rogers NH, Perfield JW 2nd, Strissel KJ, Obin MS, Greenberg AS. Reduced energy expenditure and increased inflammation are early events in the development of ovariectomy-induced obesity. Endocrinology. 2009 May;150(5):2161-8. doi: 10.1210/en.2008-1405. Epub 2009 Jan 29. PMID 19179442
- [Background] Grove KL, Fried SK, Greenberg AS, Xiao XQ, Clegg DJ. A microarray analysis of sexual dimorphism of adipose tissues in high-fat-diet-induced obese mice. Int J Obes (Lond). 2010 Jun;34(6):989-1000. doi: 10.1038/ijo.2010.12. Epub 2010 Feb 16. PMID 20157318
- [Background] Sparks LM, Ukropcova B, Smith J, Pasarica M, Hymel D, Xie H, Bray GA, Miles JM, Smith SR. Relation of adipose tissue to metabolic flexibility. Diabetes Res Clin Pract. 2009 Jan;83(1):32-43. doi: 10.1016/j.diabres.2008.09.052. Epub 2008 Nov 26. PMID 19038471
- [Background] Hirosumi J, Tuncman G, Chang L, Gorgun CZ, Uysal KT, Maeda K, Karin M, Hotamisligil GS. A central role for JNK in obesity and insulin resistance. Nature. 2002 Nov 21;420(6913):333-6. doi: 10.1038/nature01137. PMID 12447443
- [Background] Hotamisligil GS, Murray DL, Choy LN, Spiegelman BM. Tumor necrosis factor alpha inhibits signaling from the insulin receptor. Proc Natl Acad Sci U S A. 1994 May 24;91(11):4854-8. doi: 10.1073/pnas.91.11.4854. PMID 8197147
- [Background] Arkan MC, Hevener AL, Greten FR, Maeda S, Li ZW, Long JM, Wynshaw-Boris A, Poli G, Olefsky J, Karin M. IKK-beta links inflammation to obesity-induced insulin resistance. Nat Med. 2005 Feb;11(2):191-8. doi: 10.1038/nm1185. Epub 2005 Jan 30. PMID 15685170
- [Background] Macotela Y, Boucher J, Tran TT, Kahn CR. Sex and depot differences in adipocyte insulin sensitivity and glucose metabolism. Diabetes. 2009 Apr;58(4):803-12. doi: 10.2337/db08-1054. Epub 2009 Jan 9. PMID 19136652
- [Background] Guerre-Millo M, Leturque A, Girard J, Lavau M. Increased insulin sensitivity and responsiveness of glucose metabolism in adipocytes from female versus male rats. J Clin Invest. 1985 Jul;76(1):109-16. doi: 10.1172/JCI111932. PMID 3894416
- [Background] D'Eon TM, Souza SC, Aronovitz M, Obin MS, Fried SK, Greenberg AS. Estrogen regulation of adiposity and fuel partitioning. Evidence of genomic and non-genomic regulation of lipogenic and oxidative pathways. J Biol Chem. 2005 Oct 28;280(43):35983-91. doi: 10.1074/jbc.M507339200. Epub 2005 Aug 17. PMID 16109719
- [Background] Riant E, Waget A, Cogo H, Arnal JF, Burcelin R, Gourdy P. Estrogens protect against high-fat diet-induced insulin resistance and glucose intolerance in mice. Endocrinology. 2009 May;150(5):2109-17. doi: 10.1210/en.2008-0971. Epub 2009 Jan 22. PMID 19164473
- [Background] Gao H, Bryzgalova G, Hedman E, Khan A, Efendic S, Gustafsson JA, Dahlman-Wright K. Long-term administration of estradiol decreases expression of hepatic lipogenic genes and improves insulin sensitivity in ob/ob mice: a possible mechanism is through direct regulation of signal transducer and activator of transcription 3. Mol Endocrinol. 2006 Jun;20(6):1287-99. doi: 10.1210/me.2006-0012. Epub 2006 Apr 20. PMID 16627594
- [Background] Pasarica M, Sereda OR, Redman LM, Albarado DC, Hymel DT, Roan LE, Rood JC, Burk DH, Smith SR. Reduced adipose tissue oxygenation in human obesity: evidence for rarefaction, macrophage chemotaxis, and inflammation without an angiogenic response. Diabetes. 2009 Mar;58(3):718-25. doi: 10.2337/db08-1098. Epub 2008 Dec 15. PMID 19074987
- [Background] Khan T, Muise ES, Iyengar P, Wang ZV, Chandalia M, Abate N, Zhang BB, Bonaldo P, Chua S, Scherer PE. Metabolic dysregulation and adipose tissue fibrosis: role of collagen VI. Mol Cell Biol. 2009 Mar;29(6):1575-91. doi: 10.1128/MCB.01300-08. Epub 2008 Dec 29. PMID 19114551
- [Background] Haas E, Bhattacharya I, Brailoiu E, Damjanovic M, Brailoiu GC, Gao X, Mueller-Guerre L, Marjon NA, Gut A, Minotti R, Meyer MR, Amann K, Ammann E, Perez-Dominguez A, Genoni M, Clegg DJ, Dun NJ, Resta TC, Prossnitz ER, Barton M. Regulatory role of G protein-coupled estrogen receptor for vascular function and obesity. Circ Res. 2009 Feb 13;104(3):288-91. doi: 10.1161/CIRCRESAHA.108.190892. Epub 2009 Jan 29. PMID 19179659
- [Background] Belanger C, Luu-The V, Dupont P, Tchernof A. Adipose tissue intracrinology: potential importance of local androgen/estrogen metabolism in the regulation of adiposity. Horm Metab Res. 2002 Nov-Dec;34(11-12):737-45. doi: 10.1055/s-2002-38265. PMID 12660892
- [Background] Cleland WH, Mendelson CR, Simpson ER. Aromatase activity of membrane fractions of human adipose tissue stromal cells and adipocytes. Endocrinology. 1983 Dec;113(6):2155-60. doi: 10.1210/endo-113-6-2155. PMID 6641629
- [Background] Brasaemle DL, Dolios G, Shapiro L, Wang R. Proteomic analysis of proteins associated with lipid droplets of basal and lipolytically stimulated 3T3-L1 adipocytes. J Biol Chem. 2004 Nov 5;279(45):46835-42. doi: 10.1074/jbc.M409340200. Epub 2004 Aug 27. PMID 15337753
- [Background] Khor VK, Tong MH, Qian Y, Song WC. Gender-specific expression and mechanism of regulation of estrogen sulfotransferase in adipose tissues of the mouse. Endocrinology. 2008 Nov;149(11):5440-8. doi: 10.1210/en.2008-0271. Epub 2008 Jul 31. PMID 18669602
- [Background] Marin P, Krotkiewski M, Bjorntorp P. Androgen treatment of middle-aged, obese men: effects on metabolism, muscle and adipose tissues. Eur J Med. 1992 Oct;1(6):329-36. PMID 1341460
- [Background] Lovejoy JC, Champagne CM, de Jonge L, Xie H, Smith SR. Increased visceral fat and decreased energy expenditure during the menopausal transition. Int J Obes (Lond). 2008 Jun;32(6):949-58. doi: 10.1038/ijo.2008.25. Epub 2008 Mar 11. PMID 18332882
- [Background] van Nas A, Guhathakurta D, Wang SS, Yehya N, Horvath S, Zhang B, Ingram-Drake L, Chaudhuri G, Schadt EE, Drake TA, Arnold AP, Lusis AJ. Elucidating the role of gonadal hormones in sexually dimorphic gene coexpression networks. Endocrinology. 2009 Mar;150(3):1235-49. doi: 10.1210/en.2008-0563. Epub 2008 Oct 30. PMID 18974276
- [Background] Guo K, Mogen J, Struzzi S, Zhang Y. Preadipocyte transplantation: an in vivo study of direct leptin signaling on adipocyte morphogenesis and cell size. Am J Physiol Regul Integr Comp Physiol. 2009 May;296(5):R1339-47. doi: 10.1152/ajpregu.90691.2008. Epub 2009 Feb 4. PMID 19193947
- [Background] Fabian MR, Sonenberg N, Filipowicz W. Regulation of mRNA translation and stability by microRNAs. Annu Rev Biochem. 2010;79:351-79. doi: 10.1146/annurev-biochem-060308-103103. PMID 20533884
- [Background] Jones ME, Thorburn AW, Britt KL, Hewitt KN, Wreford NG, Proietto J, Oz OK, Leury BJ, Robertson KM, Yao S, Simpson ER. Aromatase-deficient (ArKO) mice have a phenotype of increased adiposity. Proc Natl Acad Sci U S A. 2000 Nov 7;97(23):12735-40. doi: 10.1073/pnas.97.23.12735. PMID 11070087
- [Background] Friso S, Choi SW, Dolnikowski GG, Selhub J. A method to assess genomic DNA methylation using high-performance liquid chromatography/electrospray ionization mass spectrometry. Anal Chem. 2002 Sep 1;74(17):4526-31. doi: 10.1021/ac020050h. PMID 12236365
- [Background] Elia M, Livesey G. Energy expenditure and fuel selection in biological systems: the theory and practice of calculations based on indirect calorimetry and tracer methods. World Rev Nutr Diet. 1992;70:68-131. doi: 10.1159/000421672. No abstract available. PMID 1292242
- [Background] Freda PU, Shen W, Reyes-Vidal CM, Geer EB, Arias-Mendoza F, Gallagher D, Heymsfield SB. Skeletal muscle mass in acromegaly assessed by magnetic resonance imaging and dual-photon x-ray absorptiometry. J Clin Endocrinol Metab. 2009 Aug;94(8):2880-6. doi: 10.1210/jc.2009-0026. Epub 2009 Jun 2. PMID 19491226
- [Background] Livingstone MB, Black AE. Markers of the validity of reported energy intake. J Nutr. 2003 Mar;133 Suppl 3:895S-920S. doi: 10.1093/jn/133.3.895S. PMID 12612176
- [Background] Schoeller DA, Racette SB. A review of field techniques for the assessment of energy expenditure. J Nutr. 1990 Nov;120 Suppl 11(11 Suppl):1492-5. doi: 10.1093/jn/120.suppl_11.1492. PMID 2243294
- [Background] Gealekman O, Guseva N, Hartigan C, Apotheker S, Gorgoglione M, Gurav K, Tran KV, Straubhaar J, Nicoloro S, Czech MP, Thompson M, Perugini RA, Corvera S. Depot-specific differences and insufficient subcutaneous adipose tissue angiogenesis in human obesity. Circulation. 2011 Jan 18;123(2):186-94. doi: 10.1161/CIRCULATIONAHA.110.970145. Epub 2011 Jan 3. PMID 21200001
- [Background] Lavau M, Susini C, Knittle J, Blanchet-Hirst S, Greenwood MR. A reliable photomicrographic method to determining fat cell size and number: application to dietary obesity. Proc Soc Exp Biol Med. 1977 Nov;156(2):251-6. doi: 10.3181/00379727-156-39916. No abstract available. PMID 928396
- [Background] Adams V, Lenk K, Linke A, Lenz D, Erbs S, Sandri M, Tarnok A, Gielen S, Emmrich F, Schuler G, Hambrecht R. Increase of circulating endothelial progenitor cells in patients with coronary artery disease after exercise-induced ischemia. Arterioscler Thromb Vasc Biol. 2004 Apr;24(4):684-90. doi: 10.1161/01.ATV.0000124104.23702.a0. Epub 2004 Feb 26. PMID 14988094
- [Background] Chironi G, Walch L, Pernollet MG, Gariepy J, Levenson J, Rendu F, Simon A. Decreased number of circulating CD34+KDR+ cells in asymptomatic subjects with preclinical atherosclerosis. Atherosclerosis. 2007 Mar;191(1):115-20. doi: 10.1016/j.atherosclerosis.2006.02.041. Epub 2006 Apr 18. PMID 16620831
- [Background] Van Craenenbroeck EM, Conraads VM, Van Bockstaele DR, Haine SE, Vermeulen K, Van Tendeloo VF, Vrints CJ, Hoymans VY. Quantification of circulating endothelial progenitor cells: a methodological comparison of six flow cytometric approaches. J Immunol Methods. 2008 Mar 20;332(1-2):31-40. doi: 10.1016/j.jim.2007.12.006. Epub 2008 Jan 18. PMID 18255093
- [Derived] Divoux A, Sandor K, Bojcsuk D, Talukder A, Li X, Balint BL, Osborne TF, Smith SR. Differential open chromatin profile and transcriptomic signature define depot-specific human subcutaneous preadipocytes: primary outcomes. Clin Epigenetics. 2018 Nov 26;10(1):148. doi: 10.1186/s13148-018-0582-0. PMID 30477572
- [Derived] Divoux A, Xie H, Li JL, Karastergiou K, Perera RJ, Chang RJ, Fried SK, Smith SR. MicroRNA-196 Regulates HOX Gene Expression in Human Gluteal Adipose Tissue. Obesity (Silver Spring). 2017 Aug;25(8):1375-1383. doi: 10.1002/oby.21896. Epub 2017 Jun 25. PMID 28649807
- See also: Home site of the Translational Research Institute for Metabolism and Diabetes — http://www.TRI-MD.org